CLINICAL TRIAL: NCT01276327
Title: Bioequivalence of a Fixed Dose Combination Tablet of Linagliptin 5 mg / Pioglitazone 30 mg Compared With Its Mono-components in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Replicate Design Study With Two Treatments in Four Crossover Periods)
Brief Title: Bioequivalence of a Fixed Dose Combination Tablet Linagliptin/Pioglitazone Compared With Its Mono-components
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1264.14; 2010-022649-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Pioglitazone

ARMS (4):
- 1 Linagliptin/Pioglitazone (Test) (Experimental): Fixed-Dose-Combination-Tablet, oral administration with 240 mL water
  Interventions: Drug: Linagliptin/Pioglitazone
- 2 Linagliptin + Pioglitazone (Ref) (Experimental): Tablets, oral administration with 240 mL water for each treatment
  Interventions: Drug: Linagliptin + Pioglitazone
- 3 Linagliptin/Pioglitazone (Test) (Experimental): Fixed-Dose-Combination-Tablet, oral administration with 240 mL water
  Interventions: Drug: Linagliptin/Pioglitazone
- 4 Linagliptin + Pioglitazone (Ref) (Experimental): Tablets, oral administration with 240 mL water for each treatment
  Interventions: Drug: Linagliptin + Pioglitazone

INTERVENTIONS:
Drug: Linagliptin + Pioglitazone — Medium doses, oral administration
  Arms: 2 Linagliptin + Pioglitazone (Ref)
Drug: Linagliptin + Pioglitazone — Medium doses, oral administration
  Arms: 4 Linagliptin + Pioglitazone (Ref)
Drug: Linagliptin/Pioglitazone — Medium dose oral administration
  Arms: 1 Linagliptin/Pioglitazone (Test)
Drug: Linagliptin/Pioglitazone — Medium dose oral administration
  Arms: 3 Linagliptin/Pioglitazone (Test)

SUMMARY:
The objective of the current study is to establish the bioequivalence of linagliptin/ pioglitazone fixed dose combination tablet compared to single tablets of linagliptin and pioglitazone administered together.

ELIGIBILITY:
Inclusion criteria:

Healthy male and female subjects

Exclusion criteria:

Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1264.14.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence TRTR: Subjects received 2 single doses of the test treatment (T; Fixed-Dose-Combination-Tablet of linagliptin 5 mg and pioglitazone 30 mg) and 2 single doses of the reference treatment (R; Individual linagliptin 5mg tablet and pioglitazone 30 mg tablet) in the sequence of TRTR.
- Sequence RTRT: Subjects received 2 single doses of the test treatment (T; Fixed-Dose-Combination-Tablet of linagliptin 5 mg and pioglitazone 30 mg) and 2 single doses of the reference treatment (R; Individual linagliptin 5mg tablet and pioglitazone 30 mg tablet) in the sequence of RTRT.
Period: Overall Study
Arm/Group | Sequence TRTR | Sequence RTRT
Started | 32 | 32
Completed | 30 | 29
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: TS - The treated set included all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence TRTR | Sequence RTRT | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (8.8) | 38.0 (9.3) | 37.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: AUC0-72 of Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 hours
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: PKS - The PKS included all evaluable subjects in the treated set who had no important PV relevant to the evaluation of bioequivalence and provided at least 1 evaluable observation for a pharmacokinetic endpoint in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- FDC L5P30 (Test): Fixed-Dose-Combination-Tablet of linagliptin 5 mg and pioglitazone 30 mg, oral administration with 240 mL water after an overnight fast
- L5+P30 (Ref): Individual linagliptin 5mg tablet and pioglitazone 30 mg tablet, oral administration with 240 mL water after an overnight fast
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
nmol*h/L | 278 (20.6) | 279 (20.6)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — Bioequivalence of the FDC tablet compared with the individual tablets of linagliptin and pioglitazone administered together; Unscaled average Bioequivalence; Adjusted gMean Ratio (Test/Ref) (%) = 99.92, 90% CI 2-sided [97.11 to 102.81], Standard Error of Mean 1.02 — Geometric standard error of mean was calculated

2. Primary Outcome: Cmax of Linagliptin
Description: Maximum measured concentration of the analyte in plasma was measured. Adjusted by-treatment geometric mean and CV were reported.
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
nmol/L | 8.65 (33.3) | 9.09 (31.2)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Unscaled average Bioequivalence; Adjusted gMean Ratio (Test/Ref) (%) = 94.17, 90% CI 2-sided [89.08 to 99.55], Standard Error of Mean 1.03 — Geometric Standard error of mean was calculated

3. Primary Outcome: AUC0-tz of Pioglitazone
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
ng*h/mL | 6370 (49.3) | 8100 (41.2)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Scaled average bioequivalence (SABE); Adjusted gMean Ratio (Test/Ref) (%) = 79.99, 90% CI 2-sided [74.65 to 85.72], Standard Error of Mean 1.04 — Geometric Standard error of mean was calculated

4. Primary Outcome: Cmax of Pioglitazone
Description: Maximum concentration of the analyte in plasma was measured. Adjusted by-treatment geometric mean and CV were calculated.
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
ng/mL | 806 (58.5) | 843 (42.7)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Scaled average bioequivalence (SABE); Adjusted gMean Ratio (Test/Ref) (%) = 97.31, 90% CI 2-sided [88.90 to 106.51], Standard Error of Mean 1.06 — Geometric standard error of mean was calculated

5. Secondary Outcome: AUC0-tz for Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point for Linagliptin
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
nmol*h/L | 278 (20.6) | 279 (20.6)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Unscaled average bioequivalence; Adjusted gMean Ratio (Test/Ref) (%) = 99.92, 90% CI 2-sided [97.10 to 102.81], Standard Error of Mean 1.02 — Geometric Standard error of mean was calculated

6. Secondary Outcome: AUC0-∞ of Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 hours extrapolated to infinity (inf) for linagliptin
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
nmol*h/L | 455 (27.4) | 447 (24.5)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Unscaled average bioequivalence; Adjusted gMean Ratio (Test/Ref) (%) = 101.85, 90% CI 2-sided [98.18 to 105.67], Standard Error of Mean 1.02 — Geometric standard error of mean was calculated

7. Secondary Outcome: AUC0-∞ of Pioglitazone
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 hours extrapolated to inf for pioglitazone
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
ng*h/mL | 6580 (47.5) | 8300 (40.4)
Statistical Analysis 1: Comparison: FDC L5P30 (Test) vs L5+P30 (Ref); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Scaled average bioequivalence (SABE); Adjusted gMean Ratio (Test/Ref) (%) = 80.79, 90% CI 2-sided [75.60 to 86.34], Standard Error of Mean 1.04 — Geometric standard error of mean was calculated

8. Secondary Outcome: Tmax for Linagliptin
Description: Time from dosing to the maximum measured concentration of the analyte in plasma for Linagliptin
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
hours | 1.73 [0.667 to 6.93] | 1.50 [0.577 to 6.93]

9. Secondary Outcome: Tmax for Pioglitazone
Description: Time from dosing to the maximum measured concentration of the analyte in plasma for pioglitazone
Time Frame: 0-72 hours (measurements at baseline, 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 11, 12, 24, 48 and 72 hours)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Number analyzed (Participants) | 62 | 63
hours | 1.00 [0.667 to 5.66] | 1.50 [0.650 to 4.90]

ADVERSE EVENTS:
Time Frame: 4 days treatment period (one day for every single dose), 35 days washout between drug administrations
Description: Treated set included all subjects who were dispensed study medication and were documented to have taken at least 1 dose of any study drug. Drug administrations were separated by washout periods of at least 35 days.
Arm/Group | FDC L5P30 (Test) | L5+P30 (Ref)
Serious Adverse Events (participants affected / at risk) | 0/62 | 1/63
Other Adverse Events (participants affected / at risk) | 13/62 | 7/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDC L5P30 (Test) (N=62) | L5+P30 (Ref) (N=63)
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDC L5P30 (Test) (N=62) | L5+P30 (Ref) (N=63)
Nasopharyngitis (Infections and infestations) | 5 | 3
Headache (Nervous system disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other